CLINICAL TRIAL: NCT02427399
Title: Conducting Outreach to Improve Cervical Cancer Screening Rates Among Underscreened Patients at an Urban Community Health Center
Brief Title: Conducting Outreach to Improve Cervical Cancer Screening Rates Among Underscreened Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenway Community Health (Other)
Responsible Party: Principal Investigator, Jenny Potter, Principal Investigator, Fenway Community Health
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: Cervical Cancer Screening
Record Dates: First submitted 2015-04-07; First posted 2015-04-28 (Estimated); Results first posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Usual care / opportunistic screening (No Intervention): This group will not be contacted by the study team in any way and will receive the general standard of care at Fenway. Patient charts are reviewed by the provider and medical team shortly before a scheduled visit to determine if the patient is due for a Pap, and if so, the patient is offered a Pap during the visit or the chance to schedule one for another date. Any proactive outreach occurs infrequently and at an ad-hoc basis, but should any proactive outreach occur, the study team will not interfere.
- Letter and informational sheet (Experimental): The patients in this group will be mailed a letter at time 0. The letter will inform the patient that she is overdue for a Pap and will also contain an informational sheet about cervical cancer and Pap tests. If the patient does not contact Fenway within 1 month to schedule an appointment, an additional letter will be sent at 1 month, and similarly again at 2 months. These letters will be the same, except that letters two and three will mention that previous attempts have been made at contact. Based on best practices in the literature, the letters will be signed by the patient's primary care provider.
  Interventions: Other: Letter and informational sheet
- Email (Experimental): The same text shared in the letter will be sent as an email to the patients in this intervention group, again at time 0, 1, and 2 months, as necessary for nonresponders. The email will be sent from the provider's email account. The email will have an informational sheet attached or included in the body of the email. The emails will be sent through MyFenway, the secure, Health Insurance Portability and Accountability Act (HIPAA)-compliant patient contact system at Fenway.
  Interventions: Other: Email
- Phone (Experimental): The patient will be telephoned and informed that they are due for a Pap, and given the opportunity to schedule an appointment over the phone immediately. As per HIPAA regulations, if the patient does not answer, a voicemail will be left saying that a Fenway representative has called and request that the patient calls back, but a reason will not be given. Some, but not all of the information contained in the info sheet will be provided during the call (see phone script). The script used is consistent with the scripts used currently for patient outreach. A voicemail will still count as one outreach attempt out of three. Patients will be contacted at time 0, 1, and 2 months as necessary for nonresponders.
  Interventions: Other: Phone
- Multimodal (Experimental): The patient will be sent a letter/informational sheet at time 0. If she does not respond within one month, she will be sent an email. If she does not respond by 2 months after the start of the intervention period, she will be called. If a patient randomly selected for this group does not have an email listed, she will receive one letter and two phone calls.
  Interventions: Other: Multimodal

INTERVENTIONS:
Other: Letter and informational sheet — The patients in this group will be mailed a letter at time 0. The letter will inform the patient that she is overdue for a Pap and will also contain an informational sheet about cervical cancer and Pap tests.
  Arms: Letter and informational sheet
Other: Email — The same text shared in the letter will be sent as an email to the patients in this intervention group, again at time 0, 1, and 2 months, as necessary for nonresponders.
  Arms: Email
Other: Phone — The patient will be telephoned and informed that they are due for a Pap, and given the opportunity to schedule an appointment over the phone immediately. Patients will be contacted at time 0, 1, and 2 months as necessary for nonresponders.
  Arms: Phone
Other: Multimodal — The patient will be sent a letter/informational sheet at time 0. If she does not respond within one month, she will be sent an email. If she does not respond by 2 months after the start of the intervention period, she will be called.
  Arms: Multimodal

SUMMARY:
The purpose of this project is to determine whether outreach to HIV-negative patients who are overdue for a Pap smear at a New England urban community health center can increase cervical cancer screening rates. It additionally seeks to determine which form of outreach - via letter, email, phone, or a mixture of those modalities- is most effective among these patients.

DETAILED DESCRIPTION:
To the investigators' knowledge, this study will be the first to assess the efficacy of email in cervical cancer screening outreach in a randomized controlled trial. It will also be one of the few randomized controlled trials to directly compare different outreach media directly, as opposed to different variations within a single medium (e.g. two different types of letters). Lastly, given the unique patient demographic makeup at Fenway, including a significant number of lesbian, bisexual and transgender patients, secondary subanalyses have the potential to significantly add to the investigators' knowledge of what media work best in conducting cervical cancer screening outreach with sexual and gender minorities, who are disproportionately underscreened compared to heterosexual cis-gendered women.

ELIGIBILITY:
Inclusion Criteria:

* Female or female-to-male transgender patients with a cervix
* HIV-negative
* Medical appointment at Fenway Community Health during calendar year 2012 who have not had a Pap smear in the past 3 years (since January 2010)

Exclusion Criteria:

* HIV-positive (due to different Pap testing guidelines)
* Male-to-female transgender patients
* Patients with a history of a hysterectomy, unless specified as partial or supracervical
* Patients aged 30-64 who had a negative Pap test in the past 5 years with simultaneous negative Human papillomavirus infection (HPV) co-testing

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1100 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Potter, MD, Principal Investigator — Fenway Community Health

REFERENCES:
- [Derived] Peitzmeier SM, Khullar K, Potter J. Effectiveness of four outreach modalities to patients overdue for cervical cancer screening in the primary care setting: a randomized trial. Cancer Causes Control. 2016 Sep;27(9):1081-91. doi: 10.1007/s10552-016-0786-6. Epub 2016 Jul 22. PMID 27447961

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care / Opportunistic Screening | Letter and Informational Sheet | Email | Phone | Multimodal
Started | 220 | 220 | 220 | 220 | 220
Completed | 206 | 204 | 208 | 202 | 205
Not Completed | 14 | 16 | 12 | 18 | 15
Not completed — Protocol Violation | 14 | 16 | 12 | 18 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care / Opportunistic Screening | Letter and Informational Sheet | Email | Phone | Multimodal | Total
Number analyzed (Participants) | 206 | 204 | 208 | 202 | 205 | 1025
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (10.8) | 30.7 (11.3) | 29.7 (10.9) | 29.5 (10.3) | 29.9 (10.0) | 30.1 (10.7)
Sex/Gender, Customized [Number; unit: participants]
  Female | 190 | 195 | 197 | 188 | 193 | 963
  Trans/FTM | 16 | 9 | 11 | 14 | 12 | 62
Race/Ethnicity, Customized [Number; unit: participants]
  White | 123 | 136 | 133 | 133 | 130 | 655
  Asian | 28 | 16 | 18 | 21 | 22 | 105
  Black | 17 | 16 | 20 | 11 | 14 | 78
  Hispanic | 12 | 14 | 16 | 15 | 18 | 75
  Multiracial | 5 | 6 | 5 | 4 | 5 | 25
  Other | 16 | 11 | 11 | 11 | 14 | 63
  Unknown | 5 | 5 | 5 | 7 | 2 | 24
Insured [Number; unit: participants] | 176 | 175 | 188 | 181 | 179 | 899
Mean Number of Medical Appointments [Mean (Standard Deviation); unit: appointments] | 10.5 (21.3) | 11.8 (30.2) | 7.4 (10.7) | 9.2 (19.6) | 8.8 (16.9) | 9.5 (20.7)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Receive a Pap Test at End of Follow up
Description: The outcome will be ascertained for each patient through chart review. The effectiveness of each intervention will be assessed through a comparison of screening rates between each of the four intervention arms (letter, email, phone, letter/email/phone) and the control arm (usual care/opportunistic screening).
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care / Opportunistic Screening | Letter and Informational Sheet | Email | Phone | Multimodal
Number analyzed (Participants) | 206 | 204 | 208 | 202 | 205
Participants | 44 | 50 | 53 | 59 | 74

2. Secondary Outcome: Proportion Receiving Pap Test at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care / Opportunistic Screening | Letter and Informational Sheet | Email | Phone | Multimodal
Number analyzed (Participants) | 206 | 204 | 208 | 202 | 205
Participants | 15 | 32 | 24 | 43 | 53

3. Secondary Outcome: Proportion Receiving Pap Test at 12 Months
Description: as for outcome 1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care / Opportunistic Screening | Letter and Informational Sheet | Email | Phone | Multimodal
Number analyzed (Participants) | 206 | 204 | 208 | 202 | 205
Participants | 34 | 42 | 45 | 53 | 70

ADVERSE EVENTS:
Arm/Group | Usual Care / Opportunistic Screening | Letter and Informational Sheet | Email | Phone | Multimodal
Serious Adverse Events (participants affected / at risk) | 0/206 | 0/204 | 0/208 | 0/202 | 0/205
Other Adverse Events (participants affected / at risk) | 0/206 | 0/204 | 0/208 | 0/202 | 0/205

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No